CLINICAL TRIAL: NCT03075722
Title: The Evaluation of a Nasal Mask for the Treatment of Obstructive Sleep Apnea (OSA): Comfort & Performance Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-205
Record Dates: First submitted 2017-03-05; First posted 2017-03-09 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saturn nasal mask (Experimental): Participants to use nasal mask in-home for 7 ± 3 days
  Interventions: Device: Saturn nasal mask

INTERVENTIONS:
Device: Saturn nasal mask — Nasal mask for the treatment of obstructive sleep apnea (OSA)

SUMMARY:
This investigation is designed to evaluate the performance (treatment and leak), comfort (subjective feedback), stability (subjective feedback, leak) as well as the participant's overall acceptance of the Saturn mask amongst OSA participants. An important factor in this investigation will be the testing of our two different seal sizes on the participants (small and medium size). A total number of 15 participants who currently use nasal or nasal pillow masks will be recruited for the trial. A subset of participants have been selected based on their anthropometric measurements collected in previous trials using nasal and nasal pillow masks at this site (CIA-103). Participants from previous NZ trials may be recruited into this trial with their consent. All the participants will be recruited by WellSleep, Wellington.

Participants will use the trial mask in home for a period of 7 ± 3 days. Baseline data will be collected from the participant during the first visit, the prior 7 days of CPAP usage data will be downloaded and stored for our analysis. The participant will use the trial device on their usual CPAP/APAP setting and device for the duration of the trial.

This study will be conducted in accordance with ICH/GCP guidelines. No deviation from the protocol will be implemented without prior review and approval of the sponsor except where it may be necessary to eliminate an immediate hazard to a research participant. In such case, the deviation will be reported to the sponsor as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* AHI ≥ 5 on diagnostic night
* Prescribed a CPAP device after successful OSA diagnosis
* Existing nasal or nasal pillow mask user

Exclusion Criteria:

* Inability to give consent
* Participants who are in a coma or a decreased level of consciousness.
* Anatomical or physiological conditions making APAP therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or may think they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Comfort | Up to 7 ± 3 days in-home
  Subjective questionnaire
Stability | Up to 7 ± 3 days in-home
  Subjective questionnaire
Objective leak data | Up to 7 ± 3 days in-home
  Obtained from participant's CPAP device
Subjective measurement of leak | Up to 7 ± 3 days in-home
  Subjective questionnaire
Draft | Up to 7 ± 3 days in-home
  Subjective questionnaire
Treatment efficacy | Up to 7 ± 3 days in-home
  Obtained from participant's CPAP device
Noise | Up to 7 ± 3 days in-home
  Subjective questionnaire

SECONDARY OUTCOMES:
Preference of mask | Up to 7 ± 3 days in-home
  Subjective questionnaire
Usability | Up to 7 ± 3 days in-home
  Subjective questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Bowen Hospital, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone